CLINICAL TRIAL: NCT06607250
Title: Prospective Study on Biparametric MRI-based Multi-planar VI-RADS for Assessing Muscle Invasion in Bladder Cancer
Brief Title: Bp-MRI Based Multi-planar VI-RADS
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-SR-353
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Bladder (Urothelial, Transitional Cell) Cancer; MRI
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Bladder cancer patients
  Interventions: Radiation: MRI

INTERVENTIONS:
Radiation: MRI — All enrolled patients underwent multiparametric magnetic resonance imaging, encompassing T2-weighted imaging (T2WI) and magnetic resonance diffusion-weighted imaging (DWI), in the coronal, sagittal, and axial planes.

SUMMARY:
This study is a prospective, single-center, observational clinical trial, enrolling 100 patients with malignant bladder tumors admitted to the Department of Urology at the People's Hospital of Jiangsu Province for treatment with transurethral resection or radical cystectomy.

All enrolled patients underwent multiparametric magnetic resonance imaging, including T2-weighted imaging (T2WI) in coronal, sagittal, and axial planes and diffusion-weighted imaging (DWI) in the same planes. The Vascular Invasion- and Invasion into the Detrusor muscle Assessment and Reporting System (VI-RADS) scores were evaluated for the enrolled patients. Diagnostic thresholds for muscle-invasive bladder cancer (MIBC) were set at VI-RADS scores ≥3 and ≥4, respectively. Descriptive statistics including sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) were calculated and compared against the surgical pathology gold standard results.

This study preliminarily validates the diagnostic performance of the 3D magnetic resonance-derived VI-RADS score in the assessment of muscle-invasive bladder cancer.

ELIGIBILITY:
Inclusion Criteria

1. Patients with indications of bladder cancer from preoperative assessments;
2. Unrestricted by gender;
3. Age of 18 years or older;
4. Absence of contraindications for Magnetic Resonance Imaging (MRI);
5. Provision of informed consent for the use of personal clinical data, pathology, and imaging for research purposes.

Exclusion Criteria

1. Time lapse exceeding one month between multiplanar Bp-MRI examination and surgical intervention;
2. Compromised MRI image quality due to significant artifacts, inadequate bladder filling, or absence of identifiable lesions within the bladder;
3. Postoperative histopathology confirming non-urothelial bladder cancer;
4. Inability to undergo surgery due to severe medical conditions, including heart failure, acute myocardial infarction, and severe cardiac or pulmonary diseases, rendering the patient unable to withstand routine surgical procedures;
5. Recent surgical procedures (e.g., Transurethral Resection of Bladder Tumor, TURBT) prior to MRI examination;
6. Any conditions identified by investigators that could potentially harm subjects or impede their ability to meet the study requirements;
7. Inability to provide written informed consent for participation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected bladder tumors due to symptoms such as hematuria.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
VI-RADS score | Immediately after enrollment
  All enrolled patients underwent multiparametric MRI, which included T2WI (coronal, sagittal, axial planes) and diffusion-weighted imaging (DWI) in the coronal, sagittal, and axial planes to evaluate the VI-RADS score. A VI-RADS score of ≥3 and ≥4 were used as cutoff values for the diagnosis of MIBC.

SECONDARY OUTCOMES:
statistical analysis | 1 day
  Sensitivity, specificity in predicting muscle invasive bladder cancer.
positive predictive value (PPV), negative predictive value (NPV) | 1 day
  statistical analysis
the Receiver Operating Characteristic (ROC) curve | 1 day
  statistical analysis
statistical analysis | 1 day
  the area under the curve (AUC) of the vi-rads score in predicting muscle invasive bladder cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China